CLINICAL TRIAL: NCT03815305
Title: Effect of Centella Asiatica on Xerotic Skin in Diabetes Mellitus Type 2: a Study on N(6)-Carboxymethyl-lysine, Interleukin 1-α, Dan Superoxide Dismutase in Stratum Corneum
Brief Title: Effect of Centella Asiatica on Xerotic Skin in Diabetes Mellitus Type 2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. Lili Legiawati, SpKK(K), Principle Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 441/UN2.F1/ETIK/2018/
Record Dates: First submitted 2019-01-18; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Xerosis Cutis; Diabetes Mellitus, Type 2
Keywords: dry skin; dm type 2; centella asiatica; superoxide dismutase; AGEs CML; IL-1α
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Centella asiatica extract; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topical CA and Placebo Oral Drug (Active Comparator): Patient given 10gr 1% CA ointment and 56 pcs of placebo drug
  Interventions: Drug: Topical CA
- Petroleum Jelly and placebo oral drug (Placebo Comparator): Patient given 10gr petroleum jelly 100% topical ointment and 56 pcs of placebo drug
  Interventions: Drug: Petroleum jelly
- Centella asiatica extract and Topical CA (Experimental): Patient given 10gr 1% CA ointment and 56 pcs of drug containing CA
  Interventions: Drug: Centella Asiatica Extract

INTERVENTIONS:
Drug: Centella Asiatica Extract — centlla asiatica oral drug at 1100 mg dose
  Other Names: Oral CA
  Arms: Centella asiatica extract and Topical CA
Drug: Topical CA — 1% centella asiatica ointment
  Other Names: Centella asiatica ointment
  Arms: Topical CA and Placebo Oral Drug
Drug: Petroleum jelly — vaseline album
  Other Names: Topical Placebo
  Arms: Petroleum Jelly and placebo oral drug

SUMMARY:
The objective of this study is to evaluate the effect of Centella asiatica on hydration status of lower leg skin of DM type 2 patients by measuring SRRC and Skin Capacitance in correlation with AGEs CML, inflammation marker IL-1α, and oxidative stress SOD in stratum corneum.

DETAILED DESCRIPTION:
This ia a double blind randomized clinical trial on patients diagnosed with DM type 2 with dry skin to assess the effect of Centella asiatica (CA) on dry skin in corellation with AGEs CML, inflammation marker IL-1α, and oxidative stress SOD in stratum corneum after four weeks of treatment. Subjects are divided into three groups of treatment. The first group treated with oral CA and topical CA, second group treated with oral placebo and topical CA, and the last group treated with oral and topical placebo. The total subjects in each treatment groups are 53 subjects. The recruited subjects will be randomized to receive three different treatments, consist of 1. First group (A) will receive combination of oral CA at 2x1100 mg dose and 1% topical CA ointment. 2. Second group (B) will receive oral placebo and topical CA 1% ointment 3. Third group (C) will receive oral placebo and petroleum jelly as topical placebo The recruited subjects will still receive the prescribed treatment for DM type 2. The treatment for dry skin will be administered for 28 days. Randomization done by our supervisor using computer program (RandlistR) by assigning code number for each subjects. The procedures of treatment administration are explained below: 1. Every subject will receive 56 capsules and 10 gram of ointment to be used in 2 weeks period. Subjects will also receive explanation on how to take the drugs 2. Oral drug are taken 2 capsules (@ 550 mg) b.i.d over 12 hours. 3. The ointment is applied two times a day 15 minutes after bath time. 4. The application have to be distributed evenly on a specific 7 x 20 cms area on lower leg. All patients will be given plastic cover to determine the area. 5. The estimation of ointment applied on every leg is as much as ½ FTU or about 0,25 gram. 6. After 2 week period ended, subject will be given the same treatment at follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Diabetes Mellitus Type 2
* <60 years old by the end of the study
* suffered from dry skin on lower leg skin area, (minimum score= 3, measured using SRRC)
* agree to not use any skin care product orally or topically on lower leg skin and any other drugs (unless its part of diabetes mellitus management)
* normal ankle brachial index value ranged from 0.91-1.3

Exclusion Criteria:

* the presence of diabetic ulcer on one of patient's foot
* the presence of infection or dermatitis on the experimented foot
* the presence of severe inflammation on the experimented skin (redness score >2 or/and fissure score >2 measured by SRRC or/and total SRRC score ranged from12-16)
* estimated glomerular filtration rate value (eGFR) < 45
* impaired liver function (increased by 2x from upper limit reference for AST/ALT)

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 159 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-01-12 (Actual); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Skin Capacitance | 1 month (evaluated every 2 weeks)
  SCap measured in (AU)
Change in SOD | 1 month (evaluated every 2 weeks)
  Superoxide Dismutase (compared to total protein)
Change in IL-1α | 1 month (evaluated every 2 weeks)
  Interleukin-1α (compared to total protein)
Change in AGEs CML | 1 month (evaluated every 2 week)
  Advanced Glycation End Product, N-(Carboxymethyl)lysine (compared to total protein)
Change in SRRC | 1 month (evaluated every 2 week)
  Specified symptom sum score. Measuring dry skin using four variables (scale, roughness, redness, and cracking) in score ranged from 1 to 4 for each variable. The highest the value marks the driest skin

CONTACTS AND LOCATIONS:
Overall Officials: Suhendro Suhendro, Doctor, Study Chair — Indonesia University
Locations (1):
- Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia